CLINICAL TRIAL: NCT02690844
Title: Effectiveness of Mucolox® and Clonazepam in Treatment of Burning Mouth Syndrome
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Sponsor: University of Alberta (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1182108
Record Dates: First submitted 2016-02-16; First posted 2016-02-24 (Estimated); Last update posted 2018-05-03 (Actual); Status verified 2016-02

CONDITIONS: Burning Mouth Syndrome
MeSH Terms: conditions — Burning Mouth Syndrome | interventions — Clonazepam

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Clonazepam (Active Comparator): Clonazepam (Klonopin®) treatment arm - 1 mg clonazepam (Klonopin® tablet) TID, dissolved in mouth for 3 minutes then expectorated
  Interventions: Drug: Clonazepam
- Mucolox® alone (Placebo Comparator): Mucolox® only - 5mL Mucolox® TID, swished around mouth for 3 minutes then expectorated
  Interventions: Drug: Mucolox® alone
- Mucolox® and clonazepam (Experimental): Mucolox® and clonazepam - 1mg Clonazepam/5mL Mucolox® TID, swished around mouth for 3 minutes then expectorated.
  Interventions: Drug: Clonazepam mixed with Mucolox®

INTERVENTIONS:
Drug: Clonazepam mixed with Mucolox® — 1mg clonazepam in 5mL Mucolox® will be used TID. Mixture will be swished around mouth for 3 minutes then spat out.
  Arms: Mucolox® and clonazepam
Drug: Mucolox® alone — 5mL Mucolox® TID. Mixture swished around mouth for 3 minutes then spat out.
  Arms: Mucolox® alone
Drug: Clonazepam — 1mg Clonazepam tablet will be used TID. Tablet dissolved in mouth, swished around and then expectorated.
  Arms: Clonazepam

SUMMARY:
What affect does the use of a mucoadhesive drug delivery system (Mucolox®) compounded with clonazepam have in the treatment of burning mouth syndrome?

There are no clinical trials reported in the literature that evaluate the use of a mucoadhesive vehicle to deliver clonazepam into the oral cavity and treat burning mouth syndrome. The use of a mucoadhesive may help to increase surface contact and elicit a greater reduction in symptoms.

DETAILED DESCRIPTION:
Question:

What affect does the use of a mucoadhesive drug delivery system (Mucolox®) compounded with clonazepam have in the treatment of burning mouth syndrome?

There are no clinical trials reported in the literature that evaluate the use of a mucoadhesive vehicle to deliver clonazepam into the oral cavity and treat burning mouth syndrome. The use of a mucoadhesive may help to increase surface contact and elicit a greater reduction in symptoms.

Study Design:

Randomized, single-blind study to be performed with 3 groups (seen below in treatment arms). Randomization will be performed by computer generated randomization to randomly allocate patients. The patients are not aware of the random group allocation. The study will involve assessment at three phases, once at initial examination (baseline), once at two weeks into treatment, and a final assessment at four weeks.

Treatment Arms:

1. Clonazepam (Klonopin®) treatment arm - 1 mg clonazepam (Klonopin® tablet) TID, dissolved in mouth for 3 minutes then expectorated
2. Mucolox® only - 5mL Mucolox® TID, swished around mouth for 3 minutes then expectorated.

3. Mucolox® and clonazepam - 1mg Clonazepam/5mL Mucolox® TID, swished around mouth for 3 minutes then expectorated.

Participants - Inclusion/Exclusion Criteria:

Study is open to men and woman. Only will accept patients over the age of 18.

Prior to inclusions, patients will have to have candida infection ruled out. Laboratory examination will be performed and serum levels of iron, ferritin, folate, vitamin B12 and glucose will be measured. Any abnormalities in these levels will lead to exclusion. If the patient is using an antidepressant or anxiolytic, they must have been on it for at least 6 months with no change in dosage. Resting salivary flow rates will be measured to rule out patients with hyposalivation (<0.1ml/min).

A standardized intra and extraoral examination will be performed to rule out: lichen planus, benign migratory glossitis and any other mucosal conditions. Any clinical indication of possible contact sensitivity to dental materials will be evaluated by patch testing.

Treatment Protocol and Data Collection:

After initial standardized examination and meeting the inclusion criteria, patients will be randomly allocated to one of the 3 different groups based upon computer generated randomization.

Patients will fill out a baseline questionnaire that includes the (VAS) and the Brief Pain Inventory Scale. Patients will fill in another questionnaire (with the same questions) at two weeks and a final time at four weeks.

The visual analogue scale will be a line with 0-10 marked on it. Patient will indicate on the scale how much pain they have had in the past week by circling a number. The Brief Pain Inventory will allow us to see how the burning mouth symptoms are affecting patients' feelings and function.

Objectives and Null Hypotheses

Primary objectives of this study are as follows:

* To compare the effectiveness of clonazepam tablets vs Mucolox® alone vs Mucolox® mixed with clonazepam on reducing pain intensity reported by subjects with primary burning mouth syndrome after two and four weeks .
* To compare the effectiveness of clonazepam tablets vs Mucolox® alone vs Mucolox® mixed with clonazepam on improving patient's ability to function.

Null Hypotheses

* Mucolox ® mixed with clonazepam is equally or less effective than clonazepam tablets for reducing burning mouth pain intensity reported by subjects.
* Mucolox ® mixed with clonazepam is equally or less effective than clonazepam tablets for improving patient feelings and function reported by subjects.

Outcomes The data will be analyzed for a decrease in symptoms as well as an improvement in feelings and function of the patient by comparing baseline to two weeks and four weeks.

Visual Analogue Scale

* Burning Mouth Syndrome pain will be reported on a scale from 0-10 with 0 being no pain and 10 being the worst pain possible
* A reduction of 1 or more will be considered significant and will count as partial improvement
* A reduction to 0 will be viewed as complete improvement.

Brief Pain Inventory

• Used to assess degree of interference that burning mouth symptoms have with day-to-day activities and quality of life

Medication Dosing 3 different treatment arms will be utilized.

1. Clonazepam (Klonopin®) treatment arm - 1 mg clonazepam (Klonopin® tablet) TID, dissolved in mouth for 3 minutes then expectorated
2. Mucolox® only - 5mL Mucolox® TID, swished around mouth for 3 minutes then expectorated.

3. Mucolox® and clonazepam - 1mg Clonazepam/5mL Mucolox® TID, swished around mouth for 3 minutes then expectorated.

All treatment arms will utilize medication TID (morning, midday and night). Maximum dose of 3 mg clonazepam will be used topically per day. Patients are told to expectorate their medication after swishing it around their mouth for 3 minutes to minimize the amount of systemic absorption of clonazepam. Patients will be followed for any potential side-effects.

ELIGIBILITY:
Inclusion Criteria:

* Presence of burning mouth symptoms that cannot be attributed to any other organic cause.

Exclusion Criteria:

* Laboratory examination will be performed and serum levels of iron, ferritin, folate, vitamin B12 and glucose will be measured. Normal levels required.
* Use of anxiolytic or antidepressant for less than 6 months prior to study.
* Resting salivary flow rates less than 0.1ml/min.
* Presence of oral mucosal disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-04; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Reduction of pain as judged by visual analogue scale (0 to 10) | 4 weeks

SECONDARY OUTCOMES:
Effect on quality of life issues using the Brief Pain Inventory | 4 weeks

IPD SHARING:
Plan to Share IPD: No